CLINICAL TRIAL: NCT07272239
Title: Combined Effects of Transcutaneous Vagus Nerve Stimulation and Modified Constraint Induced Movement Therapy on Upper Extremity Function, Cognition and Quality of Life in Individual With Chronic Stroke
Brief Title: Effects of tVNS and mCIMT in Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0270 Zara Mansha
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Vagus Nerve Stimulation; Motor Function; Modified Constraint Induced Movement Therapy; Upper Limb Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Transcutaneous Vagus Nerve Stimulation and Modified Constraint Induced Movement Therapy with Routine Physical Therapy
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation; Other: Modified Constraint Induced Movement Therapy with Routine Physical Therapy
- Group B (Experimental): Modified Constraint Induced Movement Therapy with Routine Physical Therapy
  Interventions: Other: Modified Constraint Induced Movement Therapy with Routine Physical Therapy

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — Each treatment session will last one hour, conducted three times per week on alternate days for eight weeks. The session will begin with 30 minutes of routine physical therapy, which will include active and active-assisted range of motion exercises, strengthening and coordination activities, and functional task training for the upper extremity. The following 30 minutes will include concurrent tVNS and mCIMT. tVNS will be administered through surface electrodes placed on the auricular region (tragus or cymba conchae) of the ear, with stimulation parameters set at a frequency of 25 Hz, pulse width of 250 μs, and intensity adjusted to a comfortable tingling level below the pain threshold. During this period, participants will perform task-oriented activities of the affected upper limb through functional tasks such as reaching, grasping, and object manipulation. Shaping techniques will be used to progressively increase task difficulty, and a soft mitt applied to the unaffected hand.
  Arms: Group A
Other: Modified Constraint Induced Movement Therapy with Routine Physical Therapy — Participants will also receive session lasting for one hour, with 30 minutes devoted to routine physical therapy followed by 30 minutes of mCIMT. The routine physical therapy component will include range of motion exercises, stretching, strengthening, and functional movement training similar to Group A to ensure treatment uniformity. The 30-minute mCIMT intervention will consist of intensive, task-specific practice of the affected upper limb under therapist supervision, focusing on goal-oriented functional tasks and repetitive training to enhance motor performance. A shaping approach will be used to progressively increase task complexity based on individual capability, and a soft constraint applied to the unaffected limb during the session.

SUMMARY:
Stroke is a leading cause of death and disability worldwide, resulting in significant physical and cognitive impairments. Arm weakness is most common after stroke and its treatment is recognized as an area of considerable need. The functional limitations and disabilities experienced by stroke survivors, particularly in the upper limb have a profound impact on their quality of life. Current treatment for arm weakness typically comprises intensive, task-specific and repetitive rehabilitative interventions. Transcutaneous auricular vagus nerve stimulation (tVNS) is a novel noninvasive treatment for stroke that directly stimulates the peripheral auricular branch of the vagus nerve. This study determines the effects of Vagus Nerve Stimulation and Modified Constraint Induced Movement Therapy on Motor Function, Cognition, and Quality of life in chronic stroke patients.

This randomized clinical trial will be conducted at IIMCT Railway General Hospital and Al-firdous physiotherapy clinic over a duration of six months. The sample size will consist of 50 participants. Participants which meet the inclusion criteria will be taken through non-probability convenience sampling technique, which will further be randomized through online randomization tool. 25 Participants will be assigned to Group A receiving tVNS and mCIMT with routine physical therapy and 25 to Group B receiving mCIMT with routine physical therapy . Data will be collected using various assessment tools, including Fugl-Meyer Assessment-UE (FM-UE), and Nine-hole peg test (NHPT) to assess Motor function. Stroke Impact Scale (SIS) to assess QOL, Montreal cognitive assessment (MoCA) to assess cognition, and Modified Ashworth scale to assess spasticity. All participants will receive intervention 3 days a week on alternative days for 8 weeks. Pre-intervention assessments will be conducted for both groups. The effects of the interventions will be measured at pre-treatment, 4th week, and post-intervention. Data analysis will be performed by using SPSS 26 software.

Key words: Modified Constraint Induced movement Therapy, Motor function, Rehabilitation, Stroke, Transcutaneous Vagus nerve stimulation, Upper extremity.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the leading cause of adult disability. Patients with stroke suffer from neuromuscular disabilities, including impairments in motor control. Stroke survivors with hemiplegia exhibit more upper-limb (UL) than lower-limb (LL) disability. Dysfunction from upper extremity hemi paresis impairs performance of many daily activities such as dressing, bathing, self-care and writing, thus reducing functional independence. Only 5% of adults regain full arm function after stroke, and 20% regain no functional use. Restoration of full function to the stroke affected upper extremity is a major problem in rehabilitation. Hence alternative strategies are needed to reduce the long-term disabilities and functional impairment resulting from upper extremity hemi paresis.

The severity of the neurological deficits and early patterns of improvement are the two best predictors of recovery from impairments. Patients are generally thought to experience less UL motor recovery than LL motor recovery; however, this clinical belief is typically based on disability assessments rather than tests of specific motor deficits of UL and LL. Since UL function needs finer motor control than LL function, this might explain the common scenario of less variation between impairment and disability. There are several promising treatment options available for upper-limb stroke rehabilitation, such as cross education, constraint-induced movement therapy, virtual reality therapy, functional electrical stimulation, robotic therapy, anodal transcranial direct current stimulation, and motor imagery.

Unfortunately, VNS necessitates a costly, invasive surgical procedure. In the last years, transcutaneous VNS (ta-VNS) has been proposed as a noninvasive and patient friendly method to stimulate the vagus nerve, through the skin, by delivering weak electric current to the sensory afferent fibers of the auricular, thick-myelinated, branch of the vagus nerve in the outer ear. Such stimulation activates the auricular branch of the vagus nerve and, via this pathway, the nuclei of the nerve located in the brainstem, enhancing brain GABA and Noradrenaline levels, which plays a pivotal role in brain plasticity. These connections regulate the release of neuromodulators, including acetylcholine, norepinephrine, serotonin, and brain-derived neurotrophic factors, which promote cortical plasticity.

The rationale for this study lies in its potential to uncover synergistic benefits from combining these two therapies, ultimately aiming to enhance functional recovery and cognitive engagement among chronic stroke survivors, thereby improving their daily lives and reintegration into society. The exploration of effective rehabilitation strategies is crucial, as traditional therapies frequently provide limited benefits for chronic stroke patients, particularly concerning upper extremity function. This research investigates the combined effects of ta-VNS and Modified CIMT on these patients, aiming to enhance motor recovery and cognitive engagement. The findings may inform future therapeutic approaches and offer hope for improved independence and well-being among individuals affected by chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients are included in the study.
* Left sided ischemic stroke patients.
* Patients with chronic, moderate-severe upper limb hemiparesis (>6 months-2 years)
* Stable participants having a stroke severity score > 6 on National Institute of Health Stroke Scale (NIHSS).
* Montreal Cognitive Assessment (MoCA) score ≥26.

Exclusion Criteria:

* Participants who show the symptoms of global or receptive aphasia.
* Participants who have a history of significant neurological or psychiatric disorders, other than stroke, that could interfere with upper limb motor or sensory recovery.
* Modified Ashworth scale score ≥ 3 of the affected upper extremity.
* Patients who are not able to sit with or without support.
* Patients with severe apraxia, somatosensory problems.
* Resting heart rate (< 50 beats/min).
* Participants who are currently participating in another clinical trial or research study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Fugl- Meyer Assessment- UE (FM-UE) | Assessment will be done at baseline, 4th and 8th week of intervention
  The Fugl-Meyer Assessment of Upper Extremity (FMA-UE) is a reliable and valid tool for evaluating upper limb function in stroke patients. Comprising 33 items, it assesses motor function, sensory function, and joint mobility. The FMA-UE demonstrates excellent intra-rater (ICC > 0.90) and inter-rater reliability (median agreement ~77%). It correlates well with other measures, showing strong construct validity and responsiveness, making it essential for tracking recovery in rehabilitation settings.
Nine- hole peg test (NHPT) | Assessment will be done at baseline, 4th and 8th week of intervention
  The Nine-Hole Peg Test (NHPT) is a widely used assessment tool for measuring manual dexterity and fine motor skills, particularly in clinical populations such as stroke and multiple sclerosis patients. The test involves placing and removing nine pegs from a pegboard as quickly as possible, with the time taken recorded in seconds. Reliability is strong, with intraclass correlation coefficients (ICCs) ranging from 0.91 to 0.94 for individuals with stroke and 0.49 to 0.66 for healthy adults, indicating good relative reliability. Validity is supported by its ability to discriminate between varying levels of impairment and its correlation with other dexterity measures, confirming its effectiveness in clinical settings.
Montreal cognitive assessment (MoCA) | Assessment will be done at baseline, 4th and 8th week of intervention
  The Montreal Cognitive Assessment (MoCA) is a widely utilized screening tool developed by Dr. Ziad Nasreddine in 1996 to detect cognitive impairment, particularly mild cognitive impairment (MCI) and early Alzheimer's disease. The test takes about 10 minutes and evaluates multiple cognitive domains, including memory, attention, language, executive function, and visuospatial abilities. MoCA has shown high reliability (ICC = 0.92) and good internal consistency (Cronbach's alpha = 0.82). Its sensitivity for detecting MCI is 90%, with a specificity of 87% compared to the Mini-Mental State Examination (MMSE).
Stroke impact scale (SIS) | Assessment will be done at baseline, 4th and 8th week of intervention
  The Stroke Impact Scale (SIS) is a patient-reported outcome measure designed to evaluate the effects of stroke on various aspects of life, including physical, emotional, and social domains. Developed by Duncan et al. in 1999, the SIS assesses eight dimensions: strength, hand function, mobility, activities of daily living, emotion, memory, communication, and social participation. The scale produces scores ranging from 0 to 100, with higher scores indicating better function. It has demonstrated excellent reliability (Cronbach's alpha = 0.83 to 0.95) and validity in predicting quality of life post-stroke.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Assessment will be done at baseline, 4th and 8th week of intervention
  The Modified Ashworth Scale (MAS) is a widely utilized tool for assessing spasticity, particularly in patients with neurological conditions such as stroke, cerebral palsy, and multiple sclerosis. Developed in 1987 by Bohannon and Smith, the MAS enhances the original Ashworth Scale by adding a category (1+) to improve sensitivity to lower levels of muscle tone. The scale ranges from 0 (no increase in muscle tone) to 4 (rigid in flexion or extension), allowing clinicians to evaluate resistance during passive movement. The MAS demonstrates moderate to good interrater reliability, with coefficients ranging from 0.74 to 0.93, and strong intrarater reliability values between 0.84 and 0.95. Nevertheless, it shows good correlations with other measures of muscle resistance and electromyography (EMG) parameters, making the MAS a critical tool in both clinical practice and research for evaluating spasticity and guiding treatment interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Al- firdous physiotherapy clinic, Rawalpindi, Punjab Province
  - IIMCT- Railway General Hospital, Rawalpindi, Punjab Province

REFERENCES:
- [Background] Page SJ, Sisto S, Levine P, McGrath RE. Efficacy of modified constraint-induced movement therapy in chronic stroke: a single-blinded randomized controlled trial. Arch Phys Med Rehabil. 2004 Jan;85(1):14-8. doi: 10.1016/s0003-9993(03)00481-7. PMID 14970962
- [Background] Hays SA. Enhancing Rehabilitative Therapies with Vagus Nerve Stimulation. Neurotherapeutics. 2016 Apr;13(2):382-94. doi: 10.1007/s13311-015-0417-z. PMID 26671658
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- [Background] Khodaparast N, Hays SA, Sloan AM, Hulsey DR, Ruiz A, Pantoja M, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation during rehabilitative training improves forelimb strength following ischemic stroke. Neurobiol Dis. 2013 Dec;60:80-8. doi: 10.1016/j.nbd.2013.08.002. Epub 2013 Aug 15. PMID 23954448